CLINICAL TRIAL: NCT06182436
Title: Use of Virtual Reality to Improve Pain and Anxiety Management of Children During Dupilumab Injection for Atopic Dermatitis (VR-DERMA)
Brief Title: Virtual Reality for Pain Management During Dupilumab Injection
Acronym: VR-DERMA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Sylvie Le May, Principal Investigator, St. Justine's Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: VR-DERMA
Record Dates: First submitted 2023-08-17; First posted 2023-12-27 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Atopic Dermatitis; Pain; Anxiety
MeSH Terms: conditions — Dermatitis, Atopic; Pain; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Every patient (98) will be their own control (98+98=196). Allocation to either intervention or control will be randomized at first then switched at the crossover period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Virtual Reality Distraction (Experimental): The child will play with the VR device for five minutes prior to the subcutaneous injection.
  Interventions: Device: Virtual Reality Distraction
- Standard Treatment (Active Comparator): Standard care consisting of injecting dupilumab subcutaneously without any distractive measure, with the child having full knowledge of the intervention
  Interventions: Other: Standard Treatment

INTERVENTIONS:
Device: Virtual Reality Distraction — For the experimental treatment, the child will play with the VR device for five minutes prior to the subcutaneous injection to reduce pain. The VR game Dream and the Pico Neo 4 VR headset were designed by Paperplane Therapeutics for the pediatric population. Participants will be able to direct laser beams at magical elements such as trolls and crystals. Since it is a no-success game, participants can enjoy it regardless of their past video game experience.
  Arms: Virtual Reality Distraction
Other: Standard Treatment — Standard care consisting of injecting dupilumab subcutaneously without any distractive measure, with the child having full knowledge of the intervention.
  Use of any co-interventions for pain management (music, comforting, child life specialist or other) during this sequence will be documented
  Arms: Standard Treatment

SUMMARY:
The aim of this within-subject randomized study is to examine the efficacy of a VR immersive game for pain and anxiety management of children during the subcutaneous injection of dupilumab for moderate to severe atopic dermatitis. We will recruit children from 6 to 17 years.

The main research question is:

1. Does VR immersive game will generate less anxiety and pain than standard procedures, for children receiving dupilumab injection for moderate to severe atopic dermatitis?
2. Does the occurence of side effects is similar between both study groups?

Participants will be randomized according to either sequences: VR-Standard care or Standard care-VR. During the VR sequence, participants will be playing the VR immersive game during the injection. During the Standard care sequence participants will not benefit from any pain management but passive distraction tools will be offered (and documented) to children.

The investigators will take measures of pain and anxiety, using validated scales, before and after the procedures at each sequence.

DETAILED DESCRIPTION:
Background :

Atopic dermatitis is one of the most common inflammatory diseases of the skin and usually starts in early childhood.The prevalence of atopic dermatitis ranges from 15 to 20% among children and up to 10% in adults. Atopic dermatitis treatment has been revolutionized in the past years with the approval of dupilumab (Dupixent®, Sanofi) in recent years for children. Dupilumab subcutaneous injections are highly effective in our real-world setting. However, pain at the site of injection is often reported by the parents and the patients. Regardless of the site of injection or the injection device being used, the injection remains difficult mainly because of the anxiety generated before the procedure and the anticipated pain, even if the injection only lasts five seconds.

In addition, many strategies have been unsuccessfully attempted to improve the injection experience, for example numbing cream or anxiolytic administration prior to the injection. A few authors have studied the effect of Virtual Reality (VR) on procedural pain and anxiety management. Indeed, a review of the literature has yielded only three studies who used VR with burn children. One study has verified the efficacy of VR compared to standard pharmacological care in an RCT on 54 children (6 to 19 years) suffering from burn-related injuries with TBSA (Total Body Surface Area) varying from 1 to 50%. Results showed better pain control and maximum Range of Motion (ROM) of children in the VR group.

Finally, considering the lack of optimal pain and anxiety management during dupilumab subcutaneous injections for a subset of pediatric patients, and the positive effect of an immersive distraction method such as VR for painful procedures, using VR for dupilumab injections may show promising results. To our knowledge, no other studies have tested the effect of an immersive distraction such as VR for procedural pain and anxiety management in children suffering from atopic dermatitis receiving subcutaneous injections of dupilumab.

Aim of the study

The aim of this within-subject randomized clinical trial is to verify the efficacy of an immersive distraction (virtual reality) compared to the standard of care, for pain and anxiety management of children undergoing an injection of dupilumab for moderate to severe atopic dermatitis.

Hypothesis

The use of Virtual Reality (VR) as a distraction technique during dupilumab subcutaneous injections will provide better pain and anxiety management than the standard intervention alone.

Objectives

The primary objectives are as follows:

1. To determine if VR distraction is more effective than standard care to manage procedural pain of children during dupilumab subcutaneous injections.
2. To compare if VR distraction is more effective than standard care to manage procedural anxiety of children during dupilumab subcutaneous injections.

The secondary objectives are as follows:

1. To compare if, in children with atopic dermatitis receiving subcutaneous injections of dupilumab, VR distraction generates less distressing recall of procedural pain and anxiety than the standard subcutaneous injections without distraction strategies.
2. To compare the occurrence of side effects between VR distraction and no distraction strategy in the context of dupilumab subcutaneous injections.
3. To compare healthcare professionals' satisfaction levels between VR distraction and no distraction strategy in the context of dupilumab subcutaneous injections.
4. To compare children's satisfaction levels between VR distraction and no distraction strategy in the context of dupilumab subcutaneous injections.
5. To compare parents' satisfaction levels between VR distraction and no distraction strategy in the context of dupilumab subcutaneous injections.

Methods

Design

A within-subject randomized clinical trial design with randomized sequences. Given the difficulty of ensuring any blinding conditions with the nature of the experimentation, and in order to limit the interpersonal variability between participants, each child will serve as their own control, hence receiving both standard (control) and experimental treatments (VR) during two consecutive treatment visits through a randomized order.

Sample and setting

This study will consist of 98 patients with an attrition rate of 20% where each child will serve as their own control, hence receiving both standard (control) and experimental treatments during two consecutive treatment visits through a randomized order. Thus, making a total of 196 participants. Recruitment will be done through convenience sampling of patients in the dermatology department of CHU Ste-Justine, Montreal (Qc), Canada, receiving dupilumab for moderate to severe atopic dermatitis.

Study proceedings

Every participant will be randomized to either receive the control treatment or the experimental treatment in a successive order in two different visits. Each participant will receive the two treatments and act as their own control. For the control treatment, the research nurse will administrate the subcutaneous injection as prescribed without any distractive measure, as usually performed. For the experimental treatment, the child will play with the VR device for five minutes prior to the subcutaneous injection. The participant will not be aware that the purpose of the visit is to receive the subcutaneous dupilumab injection. The child will not be informed of the exact moment of the injection and will not receive notification prior to the injection to keep the maximal effect of the immersive distraction provided by the VR experience. On the next visit, the participant will receive the other treatment, in a randomized order.

Game specifications

The VR game Dream and the Pico Neo 4 VR headset were designed by Paperplane Therapeutics for the pediatric population. In the game, participants will be able to direct laser beams at magical elements such as trolls and crystals. Since it is a no-success game, participants can enjoy it regardless of their past video game experience. The game was made to minimize cybersickness and was approved by a team of healthcare professionals in pediatric care.

Study time-points and Secondary outcomes

Measures of pain with the Verbal Numerical Rating Scale (VNRS 0-10) and anxiety with the Child Fear Scale (CFS, 0-4) will be taken before the first treatment session at (T1), after the first treatment session (T2), before the second treatment session (T3), and after the second treatment session (T4). After T2 and T4, a measure of healthcare professionals' level of satisfaction via a questionnaire developed and pretested by the team will beadministered as well. Data will also be collected on the occurrence of side effects. Clinical monitoring will be performed by an independent nurse from the research team.

Measures of the primary outcomes

Pain intensity will be assessed using the Numerical Rating Scale (NRS) for children 6 years and older immediately after the procedure during each visit (T2 and T4). The NRS is an 11-item scale for pain intensity ranging from 0 to 10; 0=no pain to 10= worst pain ever felt. This scale has an established validity (Convergent validity with Faces Pain Scale-R: r = 0.75-0.93) and reliability (Test-retest using Bland-Altman agreement: -0.9 to 1.2, 95%CI) for self-reported pain intensity in children and adolescents (6 to 17 years old). Pain intensity will also be measured at T1 and T3 to establish baseline.

The level of anxiety will be assessed using the Child Fear Scale (CFS) immediately after the procedure at each visit (T2 and T4). The CFS is a self-reported measure of anxiety adapted from the adult Faces Anxiety Scale for specific use in children undergoing painful experiences. It consists of five faces ranging from 0 (no fear/anxiety) through 4 (extremely fearful/anxious). The child is asked to indicate which face shows best how he/she felt during the procedure. Test-retest reliability has been established with children aged 5 to 10 years during painful procedure (rs = 0.76) and concurrent validity with the Children Anxiety and Pain Scale (CAPS) (rs = 0.73). The CFS was chosen because of its psychometric qualities and it is a one-item self-measure of anxiety/fear. Moreover, "although fear tends to decrease with age in general, medical fears may be an exception". Also, "age-related differences in fear ratings have not been found". Further, this scale has been used with children ranging from 5 to 18 years old for procedural fear related to venipuncture and children from 11 to 13 years for fear/anxiety of vaccine.

Sample size and statistical analysis

Recruiting 98 patients being their own control will provide a total of 196 patients which is necessary to achieve 90% power to detect a mean of paired differences of 0,40 (medium effect) with an estimated standard deviation of differences of 1,00 and with a significance level (alpha) of 0,025 using a two-sided paired t-test considering a mean difference for pain of 2.0 with a standard deviation of 1.0, a mean difference for anxiety of 1.0 with a standard deviation of 1.0 and a significance level (alpha) of 0.05/2 for both components. This sample size considers an attrition rate of 20%. Comparisons will be conducted within and between subjects for the dependent variables for repeated measures. For all variables except adverse events, an analysis of variance with one within factor condition (distraction or standard care) and one between factor order will be used. The 95% confidence interval of the difference between treatment condition will be reported. All analysis will be done in intention-to-treat using a significance level of 0,05. For primary outcomes, the Bonferroni correction will be used for the multiplicity of tests. All adverse events will be described separately by treatment condition. Statistics will be performed by an independent biostatistician.

Discussion

The investigators believe that the results of this study will provide evidence-based knowledge on a non-pharmacological method for anxiety and pain management for patients with a chronic condition undergoing a long term recurrent painful and stressful treatment through innovative interventions.

ELIGIBILITY:
Inclusion Criteria:

1. between the ages of 6 to 17 years old,
2. suffering from moderate to severe atopic dermatitis and receiving or about to start subcutaneous injections of dupilumab,
3. in the presence of a consenting parent who can understand, read, and write either French or English.

Exclusion Criteria:

1. have a diagnosed cognitive impairment precluding them from playing a virtual reality game,
2. suffer from epilepsy considering the nature of the intervention,
3. cannot be in a sitting position during the procedure as the virtual reality game requires an angle of at least 30 degrees for head-tracking.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 98 (Estimated)
Dates: Start 2024-05-16 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
mean difference in pain intensity score between sequences | Immediately after the procedure on day 1 and a week later on day 2 (T2 and T4) (self-report of pain levels during the procedure).
  Pain intensity will be assessed using the Numerical Rating Scale (NRS) for children 6 years and older. The NRS is an 11-item scale for pain intensity ranging from 0 to 10; 0=no pain to 10= worst pain ever felt.
mean difference in anxiety between sequences | Immediately after the procedure on day 1 and a week later on day 2 (T2 and T4) (self-report of anxiety levels during the procedure).
  The level of anxiety will be assessed using the Child Fear Scale (CFS). It consists of five faces ranging from 0 (no fear/anxiety) through 4 (extremely fearful/anxious). The child is asked to indicate which face shows best how he/she felt during the procedure.

SECONDARY OUTCOMES:
Mean difference in cognitive, affective and sensory components of pain as well as sense of presence in VR and engagement into the game between groups | Reported immediately after the procedure on day 1 and a week later on day 2 (T2 and T4)
  Assessed using the Graphic Rating Scale (GRS) a 7-item Likert-type scale tailored for virtual reality interventions.
children's satisfaction levels | Reported immediately after the procedure on day 1 and a week later on day 2 (T2 and T4)
  Assessed using a 0 to 10 numerical scale to answer the following question as recommended by PedIMMPACT (McGrath et al., 2008): "Considering pain relief, side effects, physical recovery, and emotional recovery, how satisfied were you with the treatments you/your child received for pain?"
healthcare professionals' satisfaction levels | Reported immediately after the sequence, a week later on day 2 (T4)
  Healthcare professional's satisfaction level will be assessed using a tailored questionnaire with four choices response scale from Strongly agree to Strongly disagree for 7 items related to their level of satisfaction with the intervention and its effect on the procedure.
Occurrence of adverse events | Reported immediately after the procedure on day 1 and a week later on day 2 (T2 and T4)
  Occurrence of adverse events will be assessed and documented from enrolment until discharge.
parents' satisfaction levels | Reported immediately after the sequence a week later on day 2 (T4)
  Parents's satisfaction levels will be assessed using a tailored questionnaire with four choices response scale from Strongly agree to Strongly disagree for 7 items related to their level of satisfaction with the intervention and its effect on the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie Le May, PhD, Principal Investigator — St. Justine's Hospital
Locations (2):
- Canada (2):
  - St. Justine's Hospital, Montreal, Quebec
  - CHU Sainte-Justine, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stander S. Atopic Dermatitis. N Engl J Med. 2021 Mar 25;384(12):1136-1143. doi: 10.1056/NEJMra2023911. No abstract available. PMID 33761208
- [Background] Thibodeaux Q, Smith MP, Ly K, Beck K, Liao W, Bhutani T. A review of dupilumab in the treatment of atopic diseases. Hum Vaccin Immunother. 2019;15(9):2129-2139. doi: 10.1080/21645515.2019.1582403. Epub 2019 Mar 27. PMID 30785362
- [Background] Kamata M, Tada Y. A Literature Review of Real-World Effectiveness and Safety of Dupilumab for Atopic Dermatitis. JID Innov. 2021 Jul 30;1(3):100042. doi: 10.1016/j.xjidi.2021.100042. eCollection 2021 Sep. PMID 34909737
- [Background] Cather J, Young M, DiRuggiero DC, Tofte S, Williams L, Gonzalez T. A Review of Phase 3 Trials of Dupilumab for the Treatment of Atopic Dermatitis in Adults, Adolescents, and Children Aged 6 and Up. Dermatol Ther (Heidelb). 2022 Sep;12(9):2013-2038. doi: 10.1007/s13555-022-00778-y. Epub 2022 Aug 26. PMID 36028787
- [Background] Hoffman HG, Meyer WJ 3rd, Ramirez M, Roberts L, Seibel EJ, Atzori B, Sharar SR, Patterson DR. Feasibility of articulated arm mounted Oculus Rift Virtual Reality goggles for adjunctive pain control during occupational therapy in pediatric burn patients. Cyberpsychol Behav Soc Netw. 2014 Jun;17(6):397-401. doi: 10.1089/cyber.2014.0058. PMID 24892204
- [Background] Dascal J, Reid M, IsHak WW, Spiegel B, Recacho J, Rosen B, Danovitch I. Virtual Reality and Medical Inpatients: A Systematic Review of Randomized, Controlled Trials. Innov Clin Neurosci. 2017 Feb 1;14(1-2):14-21. eCollection 2017 Jan-Feb. PMID 28386517
- [Background] Garrett B, Taverner T, Masinde W, Gromala D, Shaw C, Negraeff M. A rapid evidence assessment of immersive virtual reality as an adjunct therapy in acute pain management in clinical practice. Clin J Pain. 2014 Dec;30(12):1089-98. doi: 10.1097/AJP.0000000000000064. PMID 24535053
- [Background] Guo C, Deng H, Yang J. Effect of virtual reality distraction on pain among patients with hand injury undergoing dressing change. J Clin Nurs. 2015 Jan;24(1-2):115-20. doi: 10.1111/jocn.12626. Epub 2014 Jun 4. PMID 24899241
- [Background] Jeffs D, Dorman D, Brown S, Files A, Graves T, Kirk E, Meredith-Neve S, Sanders J, White B, Swearingen CJ. Effect of virtual reality on adolescent pain during burn wound care. J Burn Care Res. 2014 Sep-Oct;35(5):395-408. doi: 10.1097/BCR.0000000000000019. PMID 24823326
- [Background] Dumoulin S, Bouchard S, Ellis J, Lavoie KL, Vezina MP, Charbonneau P, Tardif J, Hajjar A. A Randomized Controlled Trial on the Use of Virtual Reality for Needle-Related Procedures in Children and Adolescents in the Emergency Department. Games Health J. 2019 Aug;8(4):285-293. doi: 10.1089/g4h.2018.0111. Epub 2019 May 24. PMID 31135178
- [Background] Gold JI, Mahrer NE. Is Virtual Reality Ready for Prime Time in the Medical Space? A Randomized Control Trial of Pediatric Virtual Reality for Acute Procedural Pain Management. J Pediatr Psychol. 2018 Apr 1;43(3):266-275. doi: 10.1093/jpepsy/jsx129. PMID 29053848
- [Background] Schneider SM, Kisby CK, Flint EP. Effect of virtual reality on time perception in patients receiving chemotherapy. Support Care Cancer. 2011 Apr;19(4):555-64. doi: 10.1007/s00520-010-0852-7. Epub 2010 Mar 26. PMID 20336327
- [Background] Wiederhold MD, Gao K, Wiederhold BK. Clinical use of virtual reality distraction system to reduce anxiety and pain in dental procedures. Cyberpsychol Behav Soc Netw. 2014 Jun;17(6):359-65. doi: 10.1089/cyber.2014.0203. PMID 24892198
- [Background] Sharar SR, Carrougher GJ, Nakamura D, Hoffman HG, Blough DK, Patterson DR. Factors influencing the efficacy of virtual reality distraction analgesia during postburn physical therapy: preliminary results from 3 ongoing studies. Arch Phys Med Rehabil. 2007 Dec;88(12 Suppl 2):S43-9. doi: 10.1016/j.apmr.2007.09.004. PMID 18036981
- [Background] Schmitt YS, Hoffman HG, Blough DK, Patterson DR, Jensen MP, Soltani M, Carrougher GJ, Nakamura D, Sharar SR. A randomized, controlled trial of immersive virtual reality analgesia, during physical therapy for pediatric burns. Burns. 2011 Feb;37(1):61-8. doi: 10.1016/j.burns.2010.07.007. Epub 2010 Aug 7. PMID 20692769
- [Background] McMurtry CM, Pillai Riddell R, Taddio A, Racine N, Asmundson GJ, Noel M, Chambers CT, Shah V; HELPinKids&Adults Team. Far From "Just a Poke": Common Painful Needle Procedures and the Development of Needle Fear. Clin J Pain. 2015 Oct;31(10 Suppl):S3-11. doi: 10.1097/AJP.0000000000000272. PMID 26352920
- [Background] Noel M, Rabbitts JA, Fales J, Chorney J, Palermo TM. The influence of pain memories on children's and adolescents' post-surgical pain experience: A longitudinal dyadic analysis. Health Psychol. 2017 Oct;36(10):987-995. doi: 10.1037/hea0000530. Epub 2017 Jul 20. PMID 28726472
- [Background] Bailey B, Daoust R, Doyon-Trottier E, Dauphin-Pierre S, Gravel J. Validation and properties of the verbal numeric scale in children with acute pain. Pain. 2010 May;149(2):216-221. doi: 10.1016/j.pain.2009.12.008. Epub 2010 Feb 25. PMID 20188471
- [Background] Castarlenas E, Jensen MP, von Baeyer CL, Miro J. Psychometric Properties of the Numerical Rating Scale to Assess Self-Reported Pain Intensity in Children and Adolescents: A Systematic Review. Clin J Pain. 2017 Apr;33(4):376-383. doi: 10.1097/AJP.0000000000000406. PMID 27518484
- [Background] Miro J, Castarlenas E, Huguet A. Evidence for the use of a numerical rating scale to assess the intensity of pediatric pain. Eur J Pain. 2009 Nov;13(10):1089-95. doi: 10.1016/j.ejpain.2009.07.002. Epub 2009 Sep 1. PMID 19726211
- [Background] Tsze DS, von Baeyer CL, Pahalyants V, Dayan PS. Validity and Reliability of the Verbal Numerical Rating Scale for Children Aged 4 to 17 Years With Acute Pain. Ann Emerg Med. 2018 Jun;71(6):691-702.e3. doi: 10.1016/j.annemergmed.2017.09.009. Epub 2017 Nov 6. PMID 29107409
- [Background] McMurtry CM, Noel M, Chambers CT, McGrath PJ. Children's fear during procedural pain: preliminary investigation of the Children's Fear Scale. Health Psychol. 2011 Nov;30(6):780-8. doi: 10.1037/a0024817. Epub 2011 Aug 1. PMID 21806301
- [Background] McKinley S, Coote K, Stein-Parbury J. Development and testing of a Faces Scale for the assessment of anxiety in critically ill patients. J Adv Nurs. 2003 Jan;41(1):73-9. doi: 10.1046/j.1365-2648.2003.02508.x. PMID 12519290
- [Background] Gullone E. The development of normal fear: a century of research. Clin Psychol Rev. 2000 Jun;20(4):429-51. doi: 10.1016/s0272-7358(99)00034-3. PMID 10832548
- [Background] Bringuier S, Dadure C, Raux O, Dubois A, Picot MC, Capdevila X. The perioperative validity of the visual analog anxiety scale in children: a discriminant and useful instrument in routine clinical practice to optimize postoperative pain management. Anesth Analg. 2009 Sep;109(3):737-44. doi: 10.1213/ane.0b013e3181af00e4. PMID 19690240
- [Background] Stoltz P, Manworren RCB. Comparison of Children's Venipuncture Fear and Pain: Randomized Controlled Trial of EMLA(R) and J-Tip Needleless Injection System(R). J Pediatr Nurs. 2017 Nov-Dec;37:91-96. doi: 10.1016/j.pedn.2017.08.025. Epub 2017 Aug 18. PMID 28823623
- [Background] Lee VY, Booy R, Skinner R, Edwards KM. The effect of exercise on vaccine-related pain, anxiety and fear during HPV vaccinations in adolescents. Vaccine. 2018 May 31;36(23):3254-3259. doi: 10.1016/j.vaccine.2018.04.069. Epub 2018 Apr 27. PMID 29709446
- [Background] Hoffman HG, Rodriguez RA, Gonzalez M, Bernardy M, Pena R, Beck W, Patterson DR, Meyer WJ 3rd. Immersive Virtual Reality as an Adjunctive Non-opioid Analgesic for Pre-dominantly Latin American Children With Large Severe Burn Wounds During Burn Wound Cleaning in the Intensive Care Unit: A Pilot Study. Front Hum Neurosci. 2019 Aug 8;13:262. doi: 10.3389/fnhum.2019.00262. eCollection 2019. PMID 31440148
- [Background] McGrath PJ, Walco GA, Turk DC, Dworkin RH, Brown MT, Davidson K, Eccleston C, Finley GA, Goldschneider K, Haverkos L, Hertz SH, Ljungman G, Palermo T, Rappaport BA, Rhodes T, Schechter N, Scott J, Sethna N, Svensson OK, Stinson J, von Baeyer CL, Walker L, Weisman S, White RE, Zajicek A, Zeltzer L; PedIMMPACT. Core outcome domains and measures for pediatric acute and chronic/recurrent pain clinical trials: PedIMMPACT recommendations. J Pain. 2008 Sep;9(9):771-83. doi: 10.1016/j.jpain.2008.04.007. Epub 2008 Jun 17. PMID 18562251
- [Background] Tesler MD, Savedra MC, Holzemer WL, Wilkie DJ, Ward JA, Paul SM. The word-graphic rating scale as a measure of children's and adolescents' pain intensity. Res Nurs Health. 1991 Oct;14(5):361-71. doi: 10.1002/nur.4770140507. PMID 1891622
- [Background] Price DD, Bush FM, Long S, Harkins SW. A comparison of pain measurement characteristics of mechanical visual analogue and simple numerical rating scales. Pain. 1994 Feb;56(2):217-226. doi: 10.1016/0304-3959(94)90097-3. PMID 8008411